CLINICAL TRIAL: NCT07016360
Title: Comparison of Efficacy of Topical Adapalene Gel Versus Cryotherapy in Recurrent Plantar Warts
Brief Title: Comparison of Effectiveness of Topical Retinoids Versus Liquid Nitrogen in Treatment of Plantar Warts(Viral Infection)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Saba Naz, DOCTOR, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192/DME/KMC
Record Dates: First submitted 2025-05-21; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Viral Warts
Keywords: Plantar warts; Topical adapalene gel; Cryotherapy
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Treated with Topical adapalene gel 0.1%
  Interventions: Drug: Topical Adapalene Gel 0.1%
- B (Experimental): Treated with liquid nitrogen over affected parts
  Interventions: Procedure: Topical Liquid Nitrogen application

INTERVENTIONS:
Drug: Topical Adapalene Gel 0.1% — Topical adapalene is a retinoid that helps in epidermal changes. Cryotherapy is a liquid nitrogen applied to affected parts for 6 months
  Arms: A
Procedure: Topical Liquid Nitrogen application — Liquid Nitrogen will be applied to affected parts.
  Arms: B

SUMMARY:
This is a comparative study between two treatment options for skin viral infection.

DETAILED DESCRIPTION:
This is a comparative study between two treatment for viral infection in epidermal layer of skin that proliferates slowly forming thick, growths. This study will compare and evaluate the differences in efficacy between topical liquid nitrogen and topical retinoids.

ELIGIBILITY:
Inclusion Criteria:

-

Patients age limit 18-60 Years Patients with either gender (Male/Female) Patients with recurrent plantar warts

Exclusion Criteria:

* Pregnancy/lactation. Pt on topical or systemic therapy in last 6 months. On immunosuppressants. > 5 lesions. Pts with local secondary infections.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Treatment | 06 months
  It will be defined through visual inspection by observing the complete clearance of the warts after 8 weeks administration of the treatment in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Saba Naz, MBBS, Principal Investigator — Khyber Teaching Hospital
Locations (1):
- Khyber Teaching Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient's confidentiality may be breached